CLINICAL TRIAL: NCT04746014
Title: Clearblue Pregnancy Test Lay User Usage Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1133
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy
Keywords: Lay User

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Clearblue Pregnancy Test — Urine Pregnancy Test

SUMMARY:
The Clearblue home pregnancy test (HPT) is an over the counter urine hCG (human chorionic gonadotrophin) visual pregnancy test which is intended for the detection of pregnancy. This study will assess the performance of the HPT in the hands of the lay user by comparing their results when used according to the instructions for use (IFU) to (i) confirmed pregnancy status of the volunteers and (ii) to the results of trained study staff testing the same urine samples.

DETAILED DESCRIPTION:
The Clearblue HPT is an over the counter urine hCG visual-read test which is intended for the detection of pregnancy. This study aims to demonstrate that the pregnancy test has the required performance characteristics in lay user testing. The study will recruit a cross-section of the target pregnancy test user population, that is, women aged over 18 years representative of the intended user.

A minimum of 300 women will be required to complete the study consisting of both pregnant and not pregnant volunteers. Each volunteer will conduct the pregnancy test using their preferred sampling method (either 'in-stream' or 'dip'). Volunteers will be evaluated against confirmed pregnancy status. Lay user comprehension of the device instructions and usability of the device will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 and over
* Interested in conducting a personal pregnancy test to determine or confirm their pregnancy status
* Willing to reveal their pregnancy status
* Willing to provide a blood sample
* Willing to give informed consent

Exclusion Criteria:

* Significant affiliation with SPD
* Used the investigational pregnancy test previously
* Qualified or trainee healthcare professional (HCP)
* Has professional experience (in current or previous job) of using dipstick type tests or lateral flow devices
* Confirmed to be pregnant by a healthcare professional and beyond the first trimester (defined as last menstrual period (LMP) +13 weeks)
* Has a medical condition that means that it is not appropriate to give a blood sample

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Study Population: Healthy pregnant or not pregnant volunteers requiring or wishing to conduct a pregnancy test to determine or confirm pregnancy status.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of Clearblue Pregnancy Test | 3 days
  Number of pregnancy tests in agreement with pregnancy status

SECONDARY OUTCOMES:
Co-ordinator Agreement | 1 day
  Number of lay users who record the same pregnancy test result as a trained study co-ordinator
Comprehension of Instructions for Use | 1 day
  Number of volunteers who answer each comprehension question correctly
Device Usability | 1 day
  Number of volunteers who record the device as easy to use

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, PhD, Study Director — SPD Development Company
Locations (1):
- WCCT, Cypress, California, United States